CLINICAL TRIAL: NCT03793361
Title: Efficacy of Regorafenib as Maintenance Therapy in Non-adipocytic Soft Tissue Sarcoma Having Received First-line Doxorubicin-based Chemotherapy
Brief Title: Phase II Study of Regorafenib as Maintenance Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EREMISS
Record Dates: First submitted 2018-12-28; First posted 2019-01-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Regorafenib
  Interventions: Drug: Regorafenib
- Arm B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regorafenib — Oral Drug in the form of 40 mg tablets - Regorafenib (120 mg/d) once daily for 3 weeks on / 1 week off plus Best Supportive Care (BSC) until progression (according to RECIST 1.1), intolerance or consent withdrawal.
  Provided by BAYER
  Other Names: stivarga
  Arms: Arm A
Drug: Placebo — Oral tablets - Placebo plus BSC until progression (according to RECIST 1.1) or unacceptable toxicity. Patients who have received placebo may be offered open-label regorafenib (cross-over option) after objective tumor progression
  Provided by BAYER
  Arms: Arm B

SUMMARY:
Multicenter double-blind placebo-controlled randomized Phase II study comparing regorafenib® to placebo, as maintenance therapy in metastatic soft-tissue non-adipocytic sarcomas experiencing stable disease or response after 6 cycles of doxorubicin-based chemotherapy as 1st line chemotherapy.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 using a centralized randomization software, assuring concealment, with a minimization program controlling for the following factors:

* Histological subgroups: leiomyosarcoma versus synovial sarcoma versus other histological subtype
* Response to doxorubicin-based chemotherapy: partial response versus stable disease
* Centers

The treatment will be administrated as long as it appears beneficial. Evaluations will be made every 8 weeks until 6 months and then every 3 months

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically proven soft tissue sarcoma including leiomyosarcoma, synovial sarcoma and other sarcomas
* Patients in partial response or stable disease after 6 cycles of doxorubicin-based first-line chemotherapy for metastatic/locally advanced soft tissue sarcoma
* Metastatic/locally advanced disease not amenable to surgical resection with curative intent
* Eastern Cooperative Oncology Group (ECOG) Performance Status =0 or 1
* Measurable disease, defined as at least 1 unidimensionally measurable lesion on a CT scan as defined by RECIST 1.1.
* Available tumor tissue for translational research program
* Adequate bone marrow, renal, and hepatic function, as evidenced by the following within 7 days of study treatment initiation:
* Absolute neutrophil count (ANC) ≥1,500/mm3
* Platelets ≥100,000/mm3
* Hemoglobin ≥9.0 g/dL
* Serum creatinine ≤1.5 x upper limit of normal (ULN)
* Glomerular filtration rate (GFR) ≥30 ml/min/1.73m2
* AST and ALT ≤2.5 x ULN ( ≤5.0 × ULN for patients with liver involvement of their cancer)
* Bilirubin ≤1.5 X ULN
* Alkaline phosphatase ≤2.5 x ULN (≤5 x ULN with liver involvement of their cancer)
* Lipase ≤1.5 x ULN
* Spot urine must not show 1+ or more protein in urine or the patient will require a repeat urine analysis. If repeat urinanalysis shows 1+ protein or more, a 24-hour urine collection will be required and must show total protein excretion <1000 mg/24 hours
* INR/PTT ≤1.5 x ULN (Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care.)
* Women of childbearing potential and male subjects must agree to use adequate contraception for the duration of study participation and up to 3 months following completion of therapy. Adequate contraception is defined as any medically recommended method (or combination of methods) as per standard of care.
* Recovery to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.0 Grade 0 or 1 level or recovery to baseline preceding the prior treatment from any previous drug/procedure related toxicity (except alopecia, anemia, and hypothyroidism).
* In the assessment of the investigator, patients are able to comply with study requirements
* Signed, IRB-approved written informed consent
* Patient covered by the French "Social Security" regime

Exclusion Criteria:

* Prior adjuvant or neoadjuvant chemotherapy not allowing at least 6 cycles of doxorubicin-based chemotherapy at metastatic stage
* Complete response to 1st line chemotherapy for metastatic/locally advanced soft tissue sarcoma
* Disease progression during the 1st line of chemotherapy
* Time interval between the last cycle of doxorubicin-based chemotherapy superior to 8 weeks
* Primary bone sarcoma
* All forms of liposarcoma
* Some particular histologic types, i.e., PNET/Ewing, alveolar or embryonal rhabdomyosarcoma, Perivascular epithelioid cell sarcoma (PECoMA), low grade endometrial stromal tumor, desmoid tumor
* Prior treatment with tyrosine kinase inhibitor
* Known history of or concomitant malignancy likely to affect life expectancy in the judgment of the investigator
* Pregnant or breastfeeding patients. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of treatment
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of Day 1 of treatment
* Active cardiac disease including any of the following: Congestive heart failure (New York Heart Association [NYHA]) ≥Class 2, Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Uncontrolled hypertension (Systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg despite optimal medical management)
* Arterial or venous thrombotic or embolic events such as myocardial infarction, cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 6 months of starting on study drug
* Any hemorrhage or bleeding event > Grade 4 within 4 weeks of start of treatment
* Ongoing infection >Grade 2 according to NCI Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v. 5.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known history of chronic hepatitis B or C
* Patients with seizure disorder requiring medication
* History of organ allograft
* Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event > Grade 4 within 4 weeks of start of treatment
* Non-healing wound, ulcer, or bone fracture
* Renal failure requiring hemo- or peritoneal dialysis
* Dehydration according to NCI-CTC v 4.0 Grade >1
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Inability to swallow oral medications, Any mal-absorption condition
* Pleural effusion or ascites that causes respiratory compromise (Grade 2 dyspnea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of regorafenib compared to placebo | from the date of randomization to the date of first observed disease progression (according to RECIST 1.1 criteria) or death from any cause, up to 12 months after the beginning of the treatment
  Progression-Free Survival will be measured from the date of randomization until the date of radiological progression (according to RECIST 1.1 criteria) or death (if death occurs before progression).

SECONDARY OUTCOMES:
To assess the efficacy of regorafenib compared to placebo | from the date of randomization to the date of death from any cause
  in terms of overall survival
To assess the efficacy of regorafenib compared to placebo | from the date of randomization to the date of first observed disease progression (according to RECIST 1.1) or death from any cause, up to 12 months after the beginning of the treatment
  Best response according to RECIST 1.1 evaluated by central radiological review: Complete Response, CR, or Partial Response, PR, achieved during the maintenance therapy. CR and PR will be counted as objective response to estimate the objective response rate (ORR)
To assess the efficacy of regorafenib compared to placebo | from the date of randomization to the date of death from any cause, up to 12 months after the beginning of the treatment
  Time to start subsequent line of anticancer therapy defined as the time interval from the date of randomization to the date of start subsequent line of anticancer therapy. Patient data will be censored at the date of last follow-up visit for patients alive at last follow-up visit without having started subsequent line of anticancer therapy. Death without having started subsequent line of anticancer therapy will be counted as a competing event.
To assess the safety of regorafenib | Baseline, every 4 weeks, up to 12 months after the beginning of the treatment
  Compared to placebo - Toxicity according to NCI-CTC AE V5.0 over the whole treatment duration plus 30 days, excluding AE unequivocally related to the disease under study or its progression. Adverse events of grade 3 or more (grade 3+) will be counted as severe adverse events
To assess the relative benefit/risk ratio | up to 12 months
  using the Q-TWiST approach - Quality-adjusted time without symptoms of disease or toxicity computed from survival times (overall survival and progression-free survival) and adverse events data (date of occurrence of grade 3+ adverse event classified as drug-related)

OTHER OUTCOMES:
assessment of the predictive value of SUMSCAN signature | up to 12 months
  genomic signature established on initial diagnostic biopsies or resection specimen and identifying sarcoma patients benefitting from anti-angiogenetic agents

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, PhD, Study Director — Centre Oscar Lambret
Locations (20):
- France (20):
  - CHRU Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Georges-François LECLERC, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital La Timone, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Institut régional du Cancer de Montpellier, Montpellier
  - Centre René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Chu Poitiers, Poitiers
  - Institut Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif